CLINICAL TRIAL: NCT05224947
Title: Gastric Layering and Monitoring II
Acronym: GLAM-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Paul Smeets, Principal Investigator, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL77717.091.21
Record Dates: First submitted 2021-12-10; First posted 2022-02-04 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Infant Formula
Keywords: Gastric behaviour; Nutrient absorption
MeSH Terms: interventions — Infant Formula

STUDY DESIGN:
Intervention Model Description: Randomized cross-over trial
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Infant formula A (Experimental)
  Interventions: Other: Infant Formula
- Infant formula B (Experimental)
  Interventions: Other: Infant Formula

INTERVENTIONS:
Other: Infant Formula — Two infant formulas differing in composition

SUMMARY:
Rationale: Results from a previous study suggest that gastric layer formation, which is caused by emulsion instability as a result of gastric acidification/digestion, is different between breastmilk and infant formula. The current study focusses on further understanding of these differences by investigating the effect of formula composition.

Objective: To investigate the effect of infant formula composition on intragastric behavior, gastric emptying and postprandial plasma parameters.

Study design: Double-blind cross-over study with two treatments.

Study population: 20 healthy normal-weight males, aged 18-45 y.

Intervention: After an overnight fast, participants will drink sufficient volume of one of the two IFs which differ in composition. Gastric content will be monitored using Magnetic Resonance Imaging (MRI). MRI scans will be done and blood samples will be taken for subsequent analyses at baseline and post prandially .

Main study parameters/endpoints: The primary outcome is gastric behavior. Secondary outcomes are total gastric content volume over time and blood parameters.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The risks associated with participation are low, as both phlebotomy and MRI are eminently safe medical techniques. In addition, the test formula are safe. Each participant will participate in 2 sessions, which require an overnight fast, 9 blood withdrawals (in total 120 mL per visit) and multiple MRI scans over a period of approximately 2 hours. These measurements are non-invasive and carry minimal risk. The burden of the sessions is most likely related to mild discomfort as they have to lie still in the MRI for two hours. This will be minimized by the soft mattress on the bed of the MRI, leg rest and a pillow underneath the head.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Apparently healthy (self-reported)
* Willing to be informed about incidental findings of pathology
* Willing to comply with the study procedures

Exclusion Criteria:

* Allergy or intolerance for cow milk, lactose, soy and/or fish (self-reported)
* Gastric disorders or regular gastric complaints, for example heart burn

  * Use of medication which alters the normal functioning of the stomach, such as: Medical drug use that influences the GI tract's normal function, e.g. motility, pH etc.: among others use of protein pump inhibitors, antacids, anti-depressants etc. (judged by study doctor)
  * Medical drug use that influences the GI tract's microbiota: antibiotic use within one month prior to the pre-study screening day (judged by study doctor)
* Smoking (>2 cigarettes a week)
* Drinking more than 14 glasses of alcohol a week
* Having given a blood donation in the past two months
* Hb value below 8.4 mmol/L (as measured with finger-prick method at screening)
* Having a contra-indication to MRI scanning, including, but not limited to:

  * Pacemakers and defibrillators
  * Intraorbital or intraocular metallic fragments
  * Ferromagnetic implants
  * Claustrophobia
* Participating in other research during the study period
* Being an employee or student of the division of human nutrition and health
* Not having a general practitioner

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Gastric layer formation over time (mL) measured with MRI | 2 hours

SECONDARY OUTCOMES:
Total gastric content volume over time (mL) | 2 hours
Concentration of glucose in blood over time | 2 hours
Concentration of insulin in blood over time | 2 hours
Concentration of free fatty acids in blood over time | 2 hours
Concentration of metabolites in blood over time measured with NMR (analysed by Nightingale: 'blood biomarker analysis service' ) | 2 hours

OTHER OUTCOMES:
Verbal ratings of hunger, fullness, bloating and nausea. | 2 hours
  Rated on a scale of 0-100, indicating 'not at all' to 'very much' respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Paul AM Smeets, PhD, Principal Investigator — Wageningen University & Research
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No